CLINICAL TRIAL: NCT02626156
Title: Monitoring and Managing Newly Healed Chronic Leg and Foot Ulcer Skin Temperature: A Cooling Intervention (MUSTCOOL) to Prevent Ulcer Recurrence
Brief Title: Cooling Leg and Foot Ulcer Skin Post Healing to Prevent Ulcer Recurrence
Acronym: MUSTCOOL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00043450
Record Dates: First submitted 2015-12-01; First posted 2015-12-10 (Estimated); Results first posted 2021-06-29 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Venous Hypertension Ulcers; Venous Stasis Ulcer; Venous Ulcer; Venous Insufficiency; Leg Ulcer; Foot Ulcer; Varicose Ulcer; Diabetic Foot
Keywords: post healed venous leg ulcer; posted healed diabetic foot ulcer
MeSH Terms: conditions — Varicose Ulcer; Venous Insufficiency; Leg Ulcer; Foot Ulcer; Diabetic Foot

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cooling gel pack (Experimental): A cooling pack will be applied to affected leg or foot skin where an ulcer has recently healed for 30 minutes three times a week (preventive maintenance). Patients will self monitor skin temperature of affected skin daily to detect elevation and will cool the affected skin daily for 5 consecutive days (bolus) if the skin temperature becomes elevated 2°F above the baseline.
  Interventions: Device: Cooling gel pack
- Cooling cotton pack (Active Comparator): A cooling cotton pack will be applied to affected leg or foot skin where an ulcer has recently healed for 30 minutes three times a week (preventive maintenance). Patients will self monitor skin temperature of affected skin daily to detect elevation and will cool the affected skin daily for 5 consecutive days (bolus) if the skin temperature becomes elevated 2°F above the baseline.
  Interventions: Device: Cooling cotton pack

INTERVENTIONS:
Device: Cooling gel pack — Individuals will self monitor skin temperature of skin over a recently health venous leg or diabetic foot ulcer with a dermal thermometer. A cooling gel pack will be applied to skin of recently healed venous leg or diabetic foot ulcers for 30 minutes 3 times a week for six months. If the temperature of this skin site increases and stays elevated 2°F above the usual temperature of that site, the individual will cool the skin 5 consecutive days and will continue to monitor skin temperature.
  Arms: Cooling gel pack
Device: Cooling cotton pack — Individuals will self monitor skin temperature of skin over a recently health venous leg or diabetic foot ulcer with a dermal thermometer. A cotton filled pack will be applied to skin of recently healed venous leg or diabetic foot ulcers for 30 minutes 3 times a week for six months. If the temperature of this skin site increases and stays elevated 2°F above the usual temperature of that site, the individual will cool the skin 5 consecutive days and will continue to monitor skin temperature.
  Arms: Cooling cotton pack

SUMMARY:
The goal of this study is to test MUSTCOOL, a home-based self-monitoring and self-management ulcer prevention intervention for patients with newly healed chronic venous leg and diabetic foot ulcers. Almost 90% of ulcers recur within 3 months of healing. During the six-month randomized clinic trial, skin temperature will be monitored daily, a maintenance dose of cooling gel pack or placebo will be applied three times weekly to the affected skin, and a bolus dose of cooling will be applied for 5 consecutive days if skin temperature becomes elevated. Outcomes on the incidence of leg ulcer recurrence, pain, physical activity and quality of life will be measured.

DETAILED DESCRIPTION:
The goal of this randomized control trial is to test a patient directed self-monitoring and self-management intervention aimed at preventing the recurrence of chronic venous leg and diabetic foot ulcers using skin temperature and cryotherapy (cooling). This MUSTCOOL study is a novel ulcer prevention strategy for patients at highest risk for developing chronic ulcers; those with a previous history. The aims are to compare a cooling treatment to a placebo to determine the outcomes on ulcer recurrence, pain, physical activity and quality of life.

Individuals with newly healed chronic ulcers will be invited to participate in MUSTCOOL's two component intervention:

1. self monitoring skin temperature over targeted "hot spots" daily with an infrared thermometer; and
2. maintenance cooling with a cooling pack (or placebo pack) placed over the "hot spot" three times each week for 30 minutes. If the temperature of the "hot spot" becomes elevated 2°F above baseline (average of 30 days of daily temperature readings) for 2 days in a row, a bolus regimen of 5 consecutive daily, 30 minute applications of the cooling or placebo pack will be implemented. The safety and side effects will be monitored, however, there have been no reported adverse events reported in our previous cryotherapy studies.

This study was designed as a chronic ulcer prevention intervention that targets the remodeling phase, the final repair process of healing after chronic ulcer closure. The skin environment is particularly vulnerable to ulcer recurrence due to a persistent aberrant inflammatory state. The previous research conducted by the study team has demonstrated that cooling this skin reduces the abnormal metabolic activity, protecting it against ulcer recurrence. Recent advancements in infrared technology allow us to take images of the affect skin to identify the area that has the highest temperature or vulnerable "hot spot". These "hot spots" will be self monitored by patients with newly healed ulcers in the home with an infrared thermometer that date and time stamps each reading. The study's outcomes on physical activity will be evaluated with an accelerometer. It is hypothesized that by improving the skin environment and reducing pain, patients will more likely be physically active and have better quality of life, all measurable goals for this study.

This prevention strategy will be evaluated over six months in 180 patients, 90 of whom will be randomized to receive the cooling pack and 90 the placebo. The goal is to test this non-pharmacological, non-invasive clinical intervention as a tailored self-management strategy to prevent chronic ulcer recurrence. It will also determine alleviation of symptoms such as pain, and the debilitating effects on physical activity and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Newly healed leg or diabetic foot ulcer within past 7 - 14 days
* Ankle brachial index 0.8- 1.3mmHg (rule out absence of arterial disease)
* Willing to wear compression stockings and appropriate footwear
* Working freezer

Exclusion Criteria:

* Open leg or foot ulcers
* Cognitive impairment: unable to recall 2 or more words or draw clock Mini-Cog™ for cognitive impairment
* Chronic inflammatory or vascular conditions where blood flow of skin may be impaired such as Lupus erythematosus, Raynaud's, scleroderma, end stage renal disease, chronic regional pain syndrome, multiple sclerosis, hypersensitivity to cold, on chemotherapy
* Unable to preform required protocol activities without assistance (return demonstration to study staff)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Moby Madisetti, MS, Study Director — Medical University of South Carolina
Locations (2):
- United States (2):
  - Medical University of South Carolina, Charleston, South Carolina
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina

REFERENCES:
- [Derived] Kelechi TJ, Mueller M, Madisetti M, Prentice M. Efficacy of a Self-managed Cooling Intervention for Pain and Physical Activity in Individuals With Recently Healed Chronic Venous Leg and Diabetic Foot Ulcers: A Randomized Controlled Trial. J Wound Ostomy Continence Nurs. 2022 Jul-Aug 01;49(4):365-372. doi: 10.1097/WON.0000000000000880. Epub 2022 May 4. PMID 35507774
- [Derived] Kelechi TJ, Madisetti M, Prentice M, Mueller M. Cooling Intervention (MUSTCOOL) for Prevention of Lower Extremity Ulcer Recurrence: A Randomized Controlled Trial. J Wound Ostomy Continence Nurs. 2021 May-Jun 01;48(3):203-210. doi: 10.1097/WON.0000000000000753. PMID 33735146

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Date recruitment period was January 2017 through December 2019 at wound clinics in the South and North Carolina areas including Charleston SC, Spartanburg SC and Greenville NC via clinicians practicing in those clinics and flyers were distributed in and around community settings such as senior centers, prior to approval from MUSC IRB.
Pre-assignment Details: 246 individuals approached, 211 prescreened eligible, 71 ineligible due to type of wound, could not make regular appointments for study visits, not interested in study, lost contact or developed infection or ulcer changed in size (healed or enlarged indicating deterioration prior to eligibility screening visit); 140 were enrolled - 58 in the DFU group (29 intervention and 29 control)and 82 in VLU group (42 intervention and 40 control)
Groups:
- Cooling Gel Pack Diabetic Foot Ulcer: A cooling pack was applied to affected foot skin where an ulcer was recently healed for 30 minutes three times a week (preventive maintenance). Participants self monitored skin temperature of affected skin daily to detect elevation and cooled the affected skin daily for 5 consecutive days (bolus) if the skin temperature became elevated 2°F above the baseline.
  Cooling gel pack: Individuals self monitored temperature of skin over a recently healed diabetic foot ulcer with a dermal thermometer. A cooling gel pack was applied to skin of recently healed diabetic foot ulcers for 30 minutes 3 times a week for six months. If the temperature of this skin site increased and stayed elevated 2°F above the usual temperature of that site, the individual cooled the skin 5 consecutive days and continued to monitor skin temperature.
- Cooling Cotton Pack Diabetic Foot Ulcer: A cooling cotton pack was applied to affected foot skin where an ulcer was recently healed, for 30 minutes three times a week (preventive maintenance). Patients self monitored temperature of affected skin daily to detect elevation and cooled the affected skin daily for 5 consecutive days (bolus) if the skin temperature became elevated 2°F above the baseline.
  Cooling cotton pack: Individuals self monitored skin temperature of skin over a recently healed diabetic foot ulcer with a dermal thermometer. A cotton filled pack was applied to skin of recently healed venous leg or diabetic foot ulcers for 30 minutes 3 times a week for six months. If the temperature of this skin site increased and stayed elevated 2°F above the usual temperature of that site, the individual cooled the skin 5 consecutive days and continued to monitor skin temperature.
- Cooling Gel Pack Venous Leg Ulcer: A cooling pack was applied to affected leg skin where an ulcer was recently healed for 30 minutes three times a week (preventive maintenance). Participants self monitored skin temperature of affected skin daily to detect elevation and cooled the affected skin daily for 5 consecutive days (bolus) if the skin temperature became elevated 2°F above the baseline.
  Cooling gel pack: Individuals self monitored temperature of skin over a recently healed venous leg or diabetic foot ulcer with a dermal thermometer. A cooling gel pack was applied to skin of recently healed venous leg ulcers for 30 minutes 3 times a week for six months. If the temperature of this skin site increased and stayed elevated 2°F above the usual temperature of that site, the individual cooled the skin 5 consecutive days and continued to monitor skin temperature.
- Cooling Cotton Pack Venous Leg Ulcer: A cooling cotton pack was applied to affected leg skin where an ulcer was recently healed, for 30 minutes three times a week (preventive maintenance). Patients self monitored temperature of affected skin daily to detect elevation and cooled the affected skin daily for 5 consecutive days (bolus) if the skin temperature became elevated 2°F above the baseline.
  Cooling cotton pack: Individuals self monitored skin temperature of skin over a recently healed venous leg ulcer with a dermal thermometer. A cotton filled pack was applied to skin of recently healed venous leg ulcers for 30 minutes 3 times a week for six months. If the temperature of this skin site increased and stayed elevated 2°F above the usual temperature of that site, the individual cooled the skin 5 consecutive days and continued to monitor skin temperature.
Period: Baseline (Visit 1 to Visit 2)
Arm/Group | Cooling Gel Pack Diabetic Foot Ulcer | Cooling Cotton Pack Diabetic Foot Ulcer | Cooling Gel Pack Venous Leg Ulcer | Cooling Cotton Pack Venous Leg Ulcer
Started | 29 | 29 | 42 | 40
Completed | 23 | 22 | 37 | 35
Not Completed | 6 | 7 | 5 | 5
Period: Study Visit 3
Arm/Group | Cooling Gel Pack Diabetic Foot Ulcer | Cooling Cotton Pack Diabetic Foot Ulcer | Cooling Gel Pack Venous Leg Ulcer | Cooling Cotton Pack Venous Leg Ulcer
Started | 23 | 22 | 37 | 35
Completed | 15 | 17 | 33 | 33
Not Completed | 8 | 5 | 4 | 2
Period: Study Visit 4
Arm/Group | Cooling Gel Pack Diabetic Foot Ulcer | Cooling Cotton Pack Diabetic Foot Ulcer | Cooling Gel Pack Venous Leg Ulcer | Cooling Cotton Pack Venous Leg Ulcer
Started | 15 | 17 | 33 | 33
Completed | 12 | 15 | 24 | 28
Not Completed | 3 | 2 | 9 | 5

BASELINE CHARACTERISTICS:
Groups:
- Cooling Gel Pack - Venous Leg Ulcer: A cooling pack was applied to affected leg skin where an ulcer was recently healed for 30 minutes three times a week (preventive maintenance). Participants self monitored skin temperature of affected skin daily to detect elevation and cooled the affected skin daily for 5 consecutive days (bolus) if the skin temperature became elevated 2°F above the baseline.
  Cooling gel pack: Individuals self monitored temperature of skin over a recently healed venous leg ulcer with a dermal thermometer. A cooling gel pack was applied to skin of recently healed venous leg ulcers for 30 minutes 3 times a week for six months. If the temperature of this skin site increased and stayed elevated 2°F above the usual temperature of that site, the individual cooled the skin 5 consecutive days and continued to monitor skin temperature.
- Cooling Cotton Pack - Venous Leg Ulcer: A cooling cotton pack was applied to affected leg skin where an ulcer was recently healed, for 30 minutes three times a week (preventive maintenance). Patients self monitored temperature of affected skin daily to detect elevation and cooled the affected skin daily for 5 consecutive days (bolus) if the skin temperature became elevated 2°F above the baseline.
  Cooling cotton pack: Individuals self monitored skin temperature of skin over a recently healed venous leg ulcer with a dermal thermometer. A cotton filled pack was applied to skin of recently healed venous leg ulcers for 30 minutes 3 times a week for six months. If the temperature of this skin site increased and stayed elevated 2°F above the usual temperature of that site, the individual cooled the skin 5 consecutive days and continued to monitor skin temperature.
- Cooling Gel Pack - Diabetic Foot Ulcer: A cooling pack was applied to affected foot skin where an ulcer was recently healed for 30 minutes three times a week (preventive maintenance). Participants self monitored skin temperature of affected skin daily to detect elevation and cooled the affected skin daily for 5 consecutive days (bolus) if the skin temperature became elevated 2°F above the baseline.
  Cooling gel pack: Individuals self monitored temperature of skin over a recently healed diabetic foot ulcer with a dermal thermometer. A cooling gel pack was applied to skin of recently healed diabetic foot ulcers for 30 minutes 3 times a week for six months. If the temperature of this skin site increased and stayed elevated 2°F above the usual temperature of that site, the individual cooled the skin 5 consecutive days and continued to monitor skin temperature.
- Cooling Cotton Pack - Diabetic Foot Ulcer: A cooling cotton pack was applied to affected foot skin where an ulcer was recently healed, for 30 minutes three times a week (preventive maintenance). Patients self monitored temperature of affected skin daily to detect elevation and cooled the affected skin daily for 5 consecutive days (bolus) if the skin temperature became elevated 2°F above the baseline.
  Cooling cotton pack: Individuals self monitored skin temperature of skin over a recently healed diabetic foot ulcer with a dermal thermometer. A cotton filled pack was applied to skin of recently healed diabetic foot ulcers for 30 minutes 3 times a week for six months. If the temperature of this skin site increased and stayed elevated 2°F above the usual temperature of that site, the individual cooled the skin 5 consecutive days and continued to monitor skin temperature.
- Total: Total of all reporting groups
Arm/Group | Cooling Gel Pack - Venous Leg Ulcer | Cooling Cotton Pack - Venous Leg Ulcer | Cooling Gel Pack - Diabetic Foot Ulcer | Cooling Cotton Pack - Diabetic Foot Ulcer | Total
Number analyzed (Participants) | 42 | 40 | 29 | 29 | 140
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (14.7) | 64.8 (12.2) | 57.8 (11.7) | 61.3 (11.6) | 62.4 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 17 | 5 | 9 | 54
  Male | 19 | 23 | 24 | 20 | 86
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3 | 1 | 7
  Not Hispanic or Latino | 39 | 40 | 26 | 28 | 133
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 20 | 14 | 8 | 5 | 47
  White | 21 | 26 | 20 | 24 | 91
  More than one race | 1 | 0 | 1 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 42 | 40 | 29 | 29 | 140

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Ulcer Recurrence
Description: Number of recurrent ulcers that develop during the 6 month study period for in participants for 4 groups of patients with previously healed venous leg ulcers receiving the cooling gel pack and cooling cotton pack and those with previously healed diabetic foot ulcers receiving the cooling gel pack or cooling cotton pack.
Time Frame: Through study completion at 6 months from baseline
Population: A total of 140 participants were randomized to either the placebo control group (n=57; 34 VLU, 23 DFU) or the intervention (n=60; 35 VLU, 25 DFU), with a final completion of 117 individuals (84%)
Measure: Number; unit: participants
Groups:
- Cotton Cooling Pack - Diabetic Foot Ulcer: A cooling cotton pack was applied to affected foot skin where an ulcer was recently healed, for 30 minutes three times a week (preventive maintenance). Patients self monitored temperature of affected skin daily to detect elevation and cooled the affected skin daily for 5 consecutive days (bolus) if the skin temperature became elevated 2°F above the baseline.
  Cooling cotton pack: Individuals self monitored skin temperature of skin over a recently healed diabetic foot ulcer with a dermal thermometer. A cotton filled pack was applied to skin of recently healed diabetic foot ulcers for 30 minutes 3 times a week for six months. If the temperature of this skin site increased and stayed elevated 2°F above the usual temperature of that site, the individual cooled the skin 5 consecutive days and continued to monitor skin temperature.
Arm/Group | Cooling Gel Pack - Venous Leg Ulcer | Cooling Cotton Pack - Venous Leg Ulcer | Cooling Gel Pack - Diabetic Foot Ulcer | Cotton Cooling Pack - Diabetic Foot Ulcer
Number analyzed (Participants) | 35 | 34 | 25 | 23
participants | 6 | 3 | 11 | 5
Statistical Analysis 1: Comparison: Cooling Gel Pack - Venous Leg Ulcer vs Cooling Cotton Pack - Venous Leg Ulcer vs Cooling Gel Pack - Diabetic Foot Ulcer vs Cotton Cooling Pack - Diabetic Foot Ulcer; Test type: Superiority; p = 0.091, Chi-squared; Risk Difference (RD) = 0.13, 95% CI 2-sided [-0.02 to 0.3], Standard Error of Mean 0.07 — Asymptotic standard error was used

2. Primary Outcome: Change in Pain (Worst Pain, Least Pain, Pain Now)
Description: Pain was measured with a visual analog scale and reported numerically (0 to 10 with 10 being the most severe pain) at baseline and at 6 months end of study
Time Frame: Through study completion at 6 months from baseline
Population: A total of 140 participants were randomized, with a final completion for this outcome of 83 individuals (59%)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Cooling Gel Pack - Venous Leg Ulcer | Cooling Cotton Pack - Venous Leg Ulcer | Cooling Gel Pack - Diabetic Foot Ulcer | Cooling Cotton Pack - Diabetic Foot Ulcer
Number analyzed (Participants) | 26 | 29 | 12 | 16
score on a scale
  Worst pain | 0.85 [-0.1 to 1.6] | 0.4 [-0.6 to 1.3] | 0 [-1.6 to 1.6] | -1.0 [-2.3 to 0.3]
  Least pain | 0.3 [-0.2 to 0.8] | 0 [-0.6 to 0.6] | -0.1 [-0.8 to 0.6] | 0 [0 to 0]
  Pain now | 0.4 [-0.06 to 0.9] | 0.14 [-0.3 to 0.5] | 0.1 [-0.1 to 0.3] | -0.1 [-0.4 to 0.1]

3. Primary Outcome: Differences in Step Counts
Description: Differences in step counts reported via accelerometer data, from baseline to post treatment at 6 months end of intervention for the 4 groups.
Time Frame: Through study completion at 6 months from baseline
Population: A total of 140 participants were randomized, with a final completion for this outcome of 75 individuals (56%)
Measure: Mean (95% Confidence Interval); unit: Steps
Arm/Group | Cooling Gel Pack - Venous Leg Ulcer | Cooling Cotton Pack - Venous Leg Ulcer | Cooling Gel Pack - Diabetic Foot Ulcer | Cotton Cooling Pack - Diabetic Foot Ulcer
Number analyzed (Participants) | 23 | 23 | 15 | 14
Steps | 17295 [9259 to 25332] | 14234 [6874 to 21593] | 13232 [2909 to 23555] | 15479 [5614 to 25343]

4. Primary Outcome: Change in Mean Scores on Quality of Life Measured With the VEINES QOL/Sym Questionnaire
Description: The Venous Insufficiency Epidemiological and Economic Study-Quality of life/Symptoms (VEINES QOL/Sym) Questionnaire was used to evaluate quality of life. A sum score is provided as an overall quality of life score for both the QOL and Sym portions of the questionnaire. This instrument was used only for the VLU groups because it is a disease-specific measure. Of the 26 items in the questionnaire, 25 items are combined to create a summary score (VEINES-QOL). One item which asks about the time of day the leg problem is most intense, question 2, provides only descriptive information and is not scored. A subset (symptoms score) of ten of these items, questions 1a to 1i and 7, is used to create a symptom score (VEINES-Sym). For both the VEINES-QOL and VEINES-Sym scores, high values indicate better outcomes. VEINES-QOL scores can be compared only to other members of the same sample. Each set of VEINES-QOL scores will have a mean T-score = 50.
Time Frame: Through study completion at 6 months from baseline
Population: Due to inadvertent scoring errors, there were data for 8 individuals.
Measure: Mean (95% Confidence Interval); unit: t-scores
Groups:
- Cooling Gel Pack: A cooling pack was applied to affected leg or foot skin where an ulcer has recently healed for 30 minutes three times a week (preventive maintenance). Patients self monitored skin temperature of affected skin daily 3 times per week to detect elevation and will cool the affected skin daily for 5 consecutive days (bolus) if the skin temperature becomes elevated 2°F above the baseline.
- Cooling Cotton Pack: A cooling cotton pack was applied to affected leg or foot skin where an ulcer has recently healed for 30 minutes three times a week (preventive maintenance). Patients self monitored skin temperature of affected skin daily to detect elevation and will cool the affected skin daily for 5 consecutive days (bolus) if the skin temperature becomes elevated 2°F above the baseline.
Arm/Group | Cooling Gel Pack | Cooling Cotton Pack
Number analyzed (Participants) | 6 | 2
t-scores
  Quality of life | 13.8 [4.0 to 23.5] | -4.8 [-121.6 to 111.9]
  Symptoms | 24.2 [13.8 to 34.5] | -4.3 [-7.4 to -1.1]

5. Primary Outcome: Changes in Severity and Intensity Pain Scores Measured With the Brief Pain Inventory
Description: The Brief Pain Inventory (BPI) scale is reported as an average score. BPI rapidly assesses the severity of pain and its impact on functioning for intensity and Pain Intensity and Pain Interference. Pain Intensity is measured in four categories: worst, least, on average, and currently, while Pain Interference is measured in 7 categories: mood, work, general activity, walking, relationships, enjoyment of life, and sleep. The patient rates each of these on a scale from 0-10, 10 being excruciating pain intensity and a complete interference in their life. Subscores are determined by averaging over the 4 intensity items for the severity subscore and over the 7 interference items for the interference subscore; possible total scores range from 0 to 10. Higher scores indicate worse intensity and severity.
Time Frame: Through study completion at 6 months from baseline
Population: A total of 140 participants were randomized, with a final completion for this outcome of 83 individuals (59%)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Cooling Gel Pack - Venous Leg Ulcer | Cooling Cotton Pack - Venous Leg Ulcer | Cooling Gel Pack - Diabetic Foot Ulcer | Cotton Cooling Pack - Diabetic Foot Ulcer
Number analyzed (Participants) | 26 | 29 | 12 | 16
score on a scale
  Severity | -0.5 [-1.0 to 0.01] | -0.2 [-0.8 to 0.4] | 0 [-0.5 to 0.5] | 0.4 [-0.1 to 0.9]
  Interference | -0.4 [-0.8 to 0.08] | -0.5 [-1.1 to 0.1] | -0.1 [-0.2 to 0.1] | 0.1 [-0.2 to 0.3]

6. Primary Outcome: Change in METS Minutes Engaging in Physical Activity Measured With The International Physical Activity Questionnaire
Description: Change in metabolic equivalent of task (METS) min per week for physical activity per The International Physical Activity Questionnaire reported for 4 groups from baseline to 6 months end of study. Scoring HIGH indicate physical activity levels equate to ~1hour of activity per day or more at least moderate intensity level or engage in vigorous intensity activity on at least 3 days achieving a minimum total physical activity of at least 1500 MET min a week or 7 or more days of any combination of walking, moderate intensity or vigorous intensity activities achieving a minimum total physical activity of at least 3000 MET min a week. MODERATE suggests engagement equivalent to 30 min of at least moderate intensity activity on most days; engage in 3 or more days of vigorous intensity activity and/or walking of at least 30 min per day or 5 or more days of moderate intensity activity and/or walking of at least 30 minutes per day. LOW level means that neither MODERATE or HIGH levels are met.
Time Frame: Through study completion at 6 months from baseline
Population: A total of 140 participants were randomized, with a final completion for this outcome of 82 individuals (59%)
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Cooling Gel Pack - Venous Leg Ulcer | Cooling Cotton Pack - Venous Leg Ulcer | Cooling Gel Pack - Diabetic Foot Ulcer | Cooling Cotton Pack - Diabetic Foot Ulcer
Number analyzed (Participants) | 25 | 29 | 12 | 16
minutes | 73 [-623 to 767] | 799 [-507 to 2104] | 1921 [1151 to 4993] | 225 [-255 to 705]

7. Primary Outcome: Time Spent in Minutes Engaging in Physical Activities
Description: Mean time spent in minutes engaging in physical activities, reported via accelerometer data, from baseline to post treatment at 6 months end of intervention for the 4 groups.
Time Frame: Through study completion at 6 months from baseline
Population: A total of 140 participants were randomized, with a final completion for this outcome of 75 individuals (56%)
Measure: Mean (95% Confidence Interval); unit: Minutes
Arm/Group | Cooling Gel Pack - Venous Leg Ulcer | Cooling Cotton Pack - Venous Leg Ulcer | Cooling Gel Pack - Diabetic Foot Ulcer | Cotton Cooling Pack - Diabetic Foot Ulcer
Number analyzed (Participants) | 23 | 23 | 15 | 14
Minutes | 1420 [-2448 to 5288] | 2523 [-765 to 5811] | 135 [28 to 242] | 157 [55 to 260]

8. Secondary Outcome: Participant Adherence to the Study Protocol
Description: Using study data logs, appropriate use of the thermometer and cooling pack was measured by the number of participants who adhered to the protocol for taking the temperature of the skin over the healed venous leg or diabetic foot ulcer. Adherence was defined as: the number of participants who were at least 80% adherent to taking their temperatures with the infrared thermometer each morning and the number of participants who were at least 80% adherent to performing the intervention every other day = 3 times times per week during the 6-month study period.
Time Frame: Daily measures starting at baseline for temperature and every other day cooling application during the 6-month study period.
Population: This outcome measured ALL participants in one group, rather than across arms, for adherence to temperature and use of cooling pack.
Measure: Count of Participants; unit: Participants
Groups:
- Adherence: All participants were assessed for adherence to the temperature and cooling protocols.
Arm/Group | Adherence
Number analyzed (Participants) | 121
Participants
  Temperature | 106
  Cooling | 82

9. Secondary Outcome: Number of Participants Indicating 'Yes' or 'Easy' on Study Instructions, Thermometer Use, Completing Logs, Performing Treatment, Helpfulness
Description: Patients satisfaction was measured by study personnel a during end of study phone survey with the following questions asked as follows (Yes/No): Were study instructions adequate, was thermometer easy to use, found cooling helpful, would cool skin area if it was proven that cooling prevented reulceration; (Easy/Not Easy): completing logs, performing the cooling treatment. Data are for (Yes/No) as number of participants who reported "yes" or if (Easy/Not Easy) the number of participants who reported "easy."
Time Frame: Survey conducted at end of the 6-month study period.
Population: A total of 140 participants were randomized, with a final completion for this outcome of 122 individuals (87%)
Measure: Number; unit: count of participants
Arm/Group | Cooling Gel Pack - Venous Leg Ulcer | Cooling Cotton Pack - Venous Leg Ulcer | Cooling Gel Pack - Diabetic Foot Ulcer | Cotton Cooling Pack - Diabetic Foot Ulcer
Number analyzed (Participants) | 36 | 34 | 27 | 25
count of participants
  Study Instructions Adequate - Yes | 36 | 34 | 26 | 25
  Using Thermometer Easy - Yes | 36 | 32 | 27 | 25
  Completing Logs - Easy | 36 | 33 | 27 | 25
  Performing Cooling -Treatment - Easy | 35 | 31 | 26 | 24
  Cooling Helpful - Yes | 31 | 21 | 21 | 18
  Would Cool if Found to Prevent Re-Ulceration - Yes | 34 | 33 | 24 | 25

10. Secondary Outcome: Knowledge Questionnaire of Study Instructions
Description: Participants were administered a 12-item (yes/no) questionnaire (test) during instruction at the start of the study, provided by the research personnel to determine comprehension of the protocol and to reinforce study procedures. Score of 12 or 100% was given for all items scoring correctly (1 point per item). Any items for which "no" was answered, remediation was conducted by study personnel at the time the questionnaire was conducted. Means scores are reported per VLU and DFU cooling pack intervention and VLU and DFU cotton cooling pack control.
Time Frame: Baseline after participant enrollment
Population: Of 140 participants, 140 (100%) completed the questionnaire.
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Cooling Cotton Pack - Venus Leg Ulcer: A cooling cotton pack was applied to affected leg skin where an ulcer was recently healed, for 30 minutes three times a week (preventive maintenance). Patients self monitored temperature of affected skin daily to detect elevation and cooled the affected skin daily for 5 consecutive days (bolus) if the skin temperature became elevated 2°F above the baseline.
  Cooling cotton pack: Individuals self monitored skin temperature of skin over a recently healed venous leg ulcer with a dermal thermometer. A cotton filled pack was applied to skin of recently healed venous leg ulcers for 30 minutes 3 times a week for six months. If the temperature of this skin site increased and stayed elevated 2°F above the usual temperature of that site, the individual cooled the skin 5 consecutive days and continued to monitor skin temperature.
- Cotton Gel Pack - Diabetic Foot Ulcer: A cooling cotton pack was applied to affected foot skin where an ulcer was recently healed, for 30 minutes three times a week (preventive maintenance). Patients self monitored temperature of affected skin daily to detect elevation and cooled the affected skin daily for 5 consecutive days (bolus) if the skin temperature became elevated 2°F above the baseline.
  Cooling cotton pack: Individuals self monitored skin temperature of skin over a recently healed diabetic foot ulcer with a dermal thermometer. A cotton filled pack was applied to skin of recently healed diabetic foot ulcers for 30 minutes 3 times a week for six months. If the temperature of this skin site increased and stayed elevated 2°F above the usual temperature of that site, the individual cooled the skin 5 consecutive days and continued to monitor skin temperature.
Arm/Group | Cooling Gel Pack - Venous Leg Ulcer | Cooling Cotton Pack - Venus Leg Ulcer | Cooling Gel Pack - Diabetic Foot Ulcer | Cotton Gel Pack - Diabetic Foot Ulcer
Number analyzed (Participants) | 42 | 40 | 29 | 29
score on a scale | 11.7 [11 to 12] | 11.9 [11 to 12] | 11.8 [11 to 12] | 11.9 [11 to 12]

ADVERSE EVENTS:
Time Frame: Data were collected for each participant for 6 months during study enrollment period.
Description: ClinicalTrial.gov definitions were used and were consistent with reporting requirements for MUSC IRB
Groups:
- Cooling Cotton Pack - Venous Leg Ulcer: A cooling cotton pack was applied to affected leg skin where an ulcer was recently healed, for 30 minutes three times a week (preventive maintenance). Patients self monitored temperature of affected skin daily to detect elevation and cooled the affected skin daily for 5 consecutive days (bolus) if the skin temperature became elevated 2°F above the baseline.
  Cooling cotton pack: Individuals self monitored skin temperature of skin over a recently healed leg ulcer with a dermal thermometer. A cotton filled pack was applied to skin of recently healed venous leg ulcers for 30 minutes 3 times a week for six months. If the temperature of this skin site increased and stayed elevated 2°F above the usual temperature of that site, the individual cooled the skin 5 consecutive days and continued to monitor skin temperature.
- Cooling Cotton Pack - Diabetic Foot Ulcer: A cooling cotton pack was applied to affected foot skin where an ulcer was recently healed, for 30 minutes three times a week (preventive maintenance). Patients self monitored temperature of affected skin daily to detect elevation and cooled the affected skin daily for 5 consecutive days (bolus) if the skin temperature became elevated 2°F above the baseline.
  Cooling cotton pack: Individuals self monitored skin temperature of skin over a recently healed foot ulcer with a dermal thermometer. A cotton filled pack was applied to skin of recently healed diabetic foot ulcers for 30 minutes 3 times a week for six months. If the temperature of this skin site increased and stayed elevated 2°F above the usual temperature of that site, the individual cooled the skin 5 consecutive days and continued to monitor skin temperature.
Arm/Group | Cooling Gel Pack - Venous Leg Ulcer | Cooling Cotton Pack - Venous Leg Ulcer | Cooling Gel Pack - Diabetic Foot Ulcer | Cooling Cotton Pack - Diabetic Foot Ulcer
All-Cause Mortality (participants affected / at risk) | 1/42 | 0/40 | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 4/42 | 2/40 | 3/29 | 4/29
Other Adverse Events (participants affected / at risk) | 14/42 | 7/40 | 15/29 | 10/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cooling Gel Pack - Venous Leg Ulcer (N=42) | Cooling Cotton Pack - Venous Leg Ulcer (N=40) | Cooling Gel Pack - Diabetic Foot Ulcer (N=29) | Cooling Cotton Pack - Diabetic Foot Ulcer (N=29)
Stroke (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Heart attack or failure (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fainted (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Amputation (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cooling Gel Pack - Venous Leg Ulcer (N=42) | Cooling Cotton Pack - Venous Leg Ulcer (N=40) | Cooling Gel Pack - Diabetic Foot Ulcer (N=29) | Cooling Cotton Pack - Diabetic Foot Ulcer (N=29)
New ulcers (Skin and subcutaneous tissue disorders) | 10 (10) | 5 (5) | 3 (3) | 4 (4) — New ulcers that developed on the treatment and non-treatment leg not involving the study healed ulcer
Recurrent ulcers (Skin and subcutaneous tissue disorders) | 6 (6) | 3 (3) | 11 (11) | 5 (5) — Recurrent ulcers of study wound
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Rash or redness of study leg or foot
Surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 3 (3) | 2 (2) — Surgeries included cataracts, orthopedic
Injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 2 (2) — Injuries from falls or other trauma
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Knee infection after surgery

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-07-23): https://cdn.clinicaltrials.gov/large-docs/56/NCT02626156/Prot_SAP_000.pdf
  • Informed Consent Form (2018-09-28): https://cdn.clinicaltrials.gov/large-docs/56/NCT02626156/ICF_001.pdf